CLINICAL TRIAL: NCT06399094
Title: Frequency-time Analysis of Pathological Lung Sounds: Detection and Quantification of Pathological Sounds in Patients With Cystic Fibrosis, Pulmonary Fibrosis or COPD (Chronic Obstructive Pulmonary Disease)
Acronym: ATF/SPP
Status: Terminated | Type: Observational
Why Stopped: Recruitment issue
Sponsor: Groupe Hospitalier de la Region de Mulhouse et Sud Alsace (Other)
Responsible Party: Sponsor
Other Study IDs: GHRMSA 1315
Record Dates: First submitted 2024-04-26; First posted 2024-05-03 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Pulmonary Fibrosis; Chronic Obstructive Pulmonary Disease; Cystic Fibrosis
MeSH Terms: conditions — Pulmonary Fibrosis; Pulmonary Disease, Chronic Obstructive; Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pulmonary fibrosis
  Interventions: Other: Lung sound recordings
- Chronic Obstructive Pulmonary Disease
  Interventions: Other: Lung sound recordings
- Cystic fibrosis
  Interventions: Other: Lung sound recordings

INTERVENTIONS:
Other: Lung sound recordings — The lung sound recordings will be made during a consultation scheduled as part of the patient's usual follow-up, after obtaining the patient's non-opposition.

SUMMARY:
The main objective of the study is to assess the potential of time-frequency representation and analysis of pulmonary sounds collected with an electronic stethoscope, as part of the routine monitoring of patients with cystic fibrosis, COPD or pulmonary fibrosis.

DETAILED DESCRIPTION:
Secondary objectives

The other objectives of this study are :

1. To evaluate the ability to detect changes in lung sounds, following optimization of the time-frequency representation.
2. To evaluate the ability to quantify differences in the severity of the pathological sounds detected using artificial intelligence and a supervised learning method.

Conduct of research This is a single-center, non-randomized, open-label study involving 60 male and female patients aged 18 to 65, eligible for a scheduled consultation as part of their usual pathological follow-up (routine care).

Lung sound recordings will be made during the same consultation, after obtaining the patient's non-opposition.

Recordings will be made using a 3M Littmann© model 3200 electronic stethoscope. The stethoscope works with Eko software, which will be installed on a touch-sensitive tablet or computer, enabling local storage of recorded data.

Whatever the patient's pathology, the physician will listen to 10 lung sites defined in the protocol. At least one breath per pulmonary site will be recorded during the consultation.

If a patient comes back for a consultation before the end of the recruitment period, a new lung sound recording will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Suffering from one of the following pathologies: cystic fibrosis, pulmonary fibrosis, COPD
* Not opposed to participating in the study

Exclusion Criteria:

* Person under court protection, guardianship or curatorship
* Person deprived of liberty by judicial or administrative decision
* Patient with a history of thoracic surgery, thoracic deformity, heart failure or other relevant illness at the investigator's discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients will be recruited during a consultation scheduled as part of the usual follow-up of their pathology in the pneumology department of mulhouse hospital center and strasbourg university hospital center.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2024-07-18 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Lung sounds visible in their representation as time-frequency images | At inclusion
  Pulmonary sounds will be recorded with an electronic stethoscope at each scheduled visit and processed with artificial intelligence using a supervised learning method.

SECONDARY OUTCOMES:
Classification of sounds by severity | At inclusion
  Pulmonary sounds will be recorded with an electronic stethoscope at each scheduled visit and processed with artificial intelligence using a supervised learning method.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpitaux Universitaire de Strasbourg, Strasbourg, Bas-Rhin
  - GHRMSA - Hôpital Emile Muller, Mulhouse, Haut-Rhin

IPD SHARING:
Plan to Share IPD: No